CLINICAL TRIAL: NCT04738370
Title: Assessment of Biomarkers in Pregnancy on Unknown Location and Ectopic Pregnancy
Acronym: ABPEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14HH2202
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy of Unknown Location; Ectopic Pregnancy; Early Pregnancy; Early Pregnancy Loss
MeSH Terms: conditions — Pregnancy, Ectopic; Abortion, Spontaneous | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (plasma and serum - plasma can assess for microRNA) +/- urine samples +/- vaginal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancy of unknown location: Patients will be approached for recruitment following PUL classification. Sample collection at time of classification +/- 48 hours later, timed for when bloods are taken as part of routine clinical practice +/- at any time patient attends for clinically indicated blood samples.
  Interventions: Other: Sample collection
- Ectopic Pregnancy: Patients will be approached for recruitment following Ectopic Pregnancy diagnosis. Ectopic pregnancies that are recruited as PUL do not need to be re-approached as they are already part of the study. Sample collection at time of diagnosis when bloods are taken as part of routine clinical practice +/- at any time patient attends for clinically indicated blood samples.
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Bloods +/- urine +/- vaginal swabs taken

SUMMARY:
To further develop the patient care pathway for women classified with a pregnancy of unknown location (PUL) and ectopic pregnancy (EP).

DETAILED DESCRIPTION:
Purpose and design-There is a need for the patient care pathway to evolve in order to aid and improve the diagnosis and management of women with a pregnancy of unknown location (PUL) and ectopic pregnancy (EP). There is potential for this to be achieved by the incorporation of a statistical model that uses one or more novel markers identified by this study.

Recruitment-1000 patients. Inclusion: Patients attending the Early Pregnancy Unit (EPU) in the first trimester with a PUL or ectopic pregnancy on trans-vaginal ultrasound scan between the ages of 18-50 years. Exclusion: Patients diagnosed with cancer, presence of acute medical condition, patients aged less than 18 years, patients who cannot give fully informed study consent.

Consent - Posters will advertise the study. Patients in EPU will be invited to the study by a member of the clinical care team. Written consent will be required.

Confidentiality - The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act. Patient consent forms will be stored securely within the study file. All patient identifiable information, where required, will be stored electronically on National Health Service (NHS) approved computers, accessible only by personnel involved in the study via password.

Conflict of interest - None involved in the study have a conflict of interest. Dissemination of results - No patient identifiable information will be included in the research report or publication. Anonymised results will be disseminated to scientific community by means of publication in peer-reviewed literature and presented at national and international meetings.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Early Pregnancy Unit in the first trimester of pregnancy (≤14 weeks gestation) aged between 18-50 years old and categorized as having a PUL or ectopic pregnancy

Exclusion Criteria:

* Younger than 18 years of age
* Women who in the opinion of the researcher by virtue of language or learning impairment would be unable to give fully informed consent to the study
* Viable intrauterine pregnancy (the presence of a fetal pole with a fetal heartbeat within the uterine cavity)
* Miscarriage
* Presence of an acute medical condition

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Pregnant women attending the Early Pregnancy Unit (EPU) within a hospital in the first trimester (up to 14 weeks gestation) with a PUL or ectopic pregnancy on trans-vaginal ultrasound scan between the ages of 18 and 50 years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-12-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PUL outcome prediction | 7 years
  The number of PUL patients correctly categorised as 'low risk' or 'high risk' based on the new logistical regression model

SECONDARY OUTCOMES:
Urinary BhCG and PUL | 7 years
  The number of PUL patients correctly categorised as 'low risk' or 'high risk' based on the interpretation of urine (rather than serum) BhCG
Urine BhCG and Ectopic pregnancy | 7 years
  The number of ectopic pregnancies correctly risk stratified as being suitable for expectant or medical management based on the interpretation of urine (rather than serum) BhCG
Plasma and Serum and PUL | 7 years
  Whether novel biomarkers present in serum and/or plasma and/or urine may have predictive value in determining 'low risk' versus 'high risk' PUL
Plasma and Serum and Ectopic pregnancy | 7 years
  Whether novel biomarkers present in serum and/or plasma and/or urine may have predictive value in determining which women diagnosed with an ectopic pregnancy are suitable for expectant or medical management
BhCG timing | 7 years
  Whether the timing of serial BhCG measurements has a significant impact on the risk stratification of PUL patients
Novel biomarkers | 7 years
  Whether a novel candidate metabolite may have predictive value in determining 'low risk' versus 'high risk' PUL
Other novel biomarkers | 7 years
  Whether a novel candidate metabolite may have predictive value in determining which women diagnosed with an ectopic pregnancy are suitable for expectant or medical management

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kyriacou C, Yang W, Kapur S, Maheetharan S, Pikovsky M, Parker N, Barcroft J, Bobdiwala S, Sur S, Stalder C, Gould D, Ofili-Yebovi D, Day A, Unsworth N, Wilkes EH, Tan T, Bourne T. Ambulatory human chorionic gonadotrophin (hCG) testing: a verification of two hCG point of care devices. Clin Chem Lab Med. 2023 Oct 30;62(4):664-673. doi: 10.1515/cclm-2023-0703. Print 2024 Mar 25. PMID 37886834